CLINICAL TRIAL: NCT05257434
Title: Postoperative Outcomes in Patients With Hepato-biliary-pancreatic Cancer According to inBody Test
Status: Recruiting | Type: Observational
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Department of Gastroenterological Surgery, Kochi University
Other Study IDs: Point study
Record Dates: First submitted 2022-02-01; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: inbody — Body fluid composition

SUMMARY:
postoperative outcomes were evaluated by using inBody test

DETAILED DESCRIPTION:
postoperative outcomes were evaluated by using inBody test

ELIGIBILITY:
Inclusion Criteria:

* surgically treated patients

Exclusion Criteria:

* a body weight loss of >10% during the 6 months before surgery; the presence of distant metastases; or seriously impaired function of vital organs because of respiratory, renal, or heart disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgically treated patients who were suffering from hepato-biliary-pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
long-term outcomes | 5year
  overall survival rate

SECONDARY OUTCOMES:
short-term outcomes | up to 24 weeks
  postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Takehiro Okabayashi, Kochi, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kimura J, Sui K, Tabuchi M, Sakamoto S, Murokawa T, Iwata J, Morita S, Iiyama T, Okabayashi T. Preoperative percent body fat in bioelectrical impedance analysis predicts pancreatic fistula after pancreaticoduodenectomy. Langenbecks Arch Surg. 2023 Jun 28;408(1):248. doi: 10.1007/s00423-023-02998-y. PMID 37380749